CLINICAL TRIAL: NCT04312542
Title: Systemic Markers of Inflammation: 9- and 12-Month Follow-Up Post Non-Surgical Periodontal Therapy With and Without Minocycline HCl Microspheres, 1mg
Brief Title: Systemic Markers of Inflammation: 9- and 12-Month Follow-Up Post Non-Surgical Periodontal Therapy
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: DENT-2020-28624
Record Dates: First submitted 2020-03-13; First posted 2020-03-18 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: SRP; Minocycline HCl Microspheres; Biomarkers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SRP with minocycline HCl microspheres: Participants in this cohort received the intervention of minocycline HCl microspheres, 1 mg in the interventional phase of the trial.
  Interventions: Procedure: Measurement of Biomarkers
- SRP without minocycline HCl microspheres: Participants in this cohort did not have minocycline HCl microspheres, 1 mg administered during the interventional phase of the trial.
  Interventions: Procedure: Measurement of Biomarkers

INTERVENTIONS:
Procedure: Measurement of Biomarkers — Participants will have blood drawn at a 9-month and 12-month visit for the measurement of biomarkers.

SUMMARY:
The primary goal of this study is to determine the amount of three systemic markers of inflammation: 1) Hemoglobin A1c (Hgb A1c, 2) High Sensitivity C-Reactive Protein (hsCRP), and 3) Haptoglobin (Hp) at 9 and 12 month follow-up post scaling and rootplaning (SRP) with and without minocycline HCl microspheres, 1 mg.

DETAILED DESCRIPTION:
Participants from a randomized controlled clinical trial approved by the University of Minnesota (UMN) Institutional Review Board (IRB) STUDY00004876 and registered on ClinicalTrials.gov (NCT03762915) identifying the effects of SRP with and without minocycline HCl microspheres, 1 mg on periodontal pathogens and systemic inflammatory markers in the blood serum will be invited to participate in this 9 and 12 month follow-up study.

ELIGIBILITY:
Inclusion Criteria:

- Participated in interventional phase of the trial STUDY00004876

Exclusion Criteria:

* Unable to comply with study protocol
* Cigarette use within the last year
* ≥2 weeks of antibiotic use in the past three months or antibiotic use in the last six weeks.
* Pregnant, planning to become pregnant, or unsure of pregnancy status (self- reported)
* Diagnosed cardiac conditions (cardiovascular disease (CVD) or atherosclerotic vascular disease (ASVD) including coronary heart disease, cerebrovascular disease, and peripheral artery disease, myocardial infarction, stroke, stable or unstable angina, transient ischemic attack, or coronary or other arterial revascularization
* Have any uncontrolled medical condition or immunocompromised that may impact the study (uncontrolled diabetes HbA1c > 7, HIV, etc.)
* Any medication that may impact periodontal conditions (Phenytoin, calciumantagonists, cyclosporin, warfarin, or NSAIDS)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants from a randomized controlled clinical trial approved by the University of Minnesota (UMN) Institutional Review Board (IRB) STUDY00004876 and registered on ClinicalTrials.gov (NCT03762915) identifying the effects of SRP with and without minocycline HCl microspheres, 1 mg on periodontal pathogens and systemic inflammatory markers in the blood serum will be invited to participate in this 9 and 12 month follow-up study.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-07-21 (Actual); Primary Completion 2022-08-16 (Actual); Study Completion 2022-08-16 (Actual)

PRIMARY OUTCOMES:
Serum Hemoglobin A1C Concentration | 9 months
  Serum hemoglobin A1C (hbA1c) concentration will be measured using enzyme-linked immunosorbant assay (ELISA) and reported in standard clinical units (percent glycolated erythrocytes).
Serum Hemoglobin A1C Concentration | 12 months
  Serum hemoglobin A1C (hbA1c) concentration will be measured using enzyme-linked immunosorbant assay (ELISA) and reported in standard clinical units (percent glycolated erythrocytes).
Serum High Sensitivity C-Reactive Protein (hsCRP) Concentration | 9 months
  Serum high sensitivity CRP concentration will be measured using enzyme-linked immunosorbant assay (ELISA) and reported in units of mg/l.
Serum High Sensitivity C-Reactive Protein (hsCRP) Concentration | 12 months
  Serum high sensitivity CRP concentration will be measured using enzyme-linked immunosorbant assay (ELISA) and reported in units of mg/l.
Serum Haptoglobin Concentration | 9 months
  Serum haptoglobin concentration will be measured using enzyme-linked immunosorbant assay (ELISA) and reported in units of mg/dl.
Serum Haptoglobin Concentration | 12 months
  Serum haptoglobin concentration will be measured using enzyme-linked immunosorbant assay (ELISA) and reported in units of mg/dl.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle B Arnett, RDH, BS, MS, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States